CLINICAL TRIAL: NCT04886726
Title: Post-transplant Cyclophosphamide and Urinary-derived Human Chorionic Gonadotropin and Epidermal Growth Factor (uhCG/EGF) as Graft Versus Host Disease Prophylaxis for Mismatched Unrelated Donor Transplantation
Brief Title: PTCY Plus uhCG/EGF for Graft Versus Host Disease Prophylaxis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Shatha Farhan, Clinical Assistant Professor, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14916
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PTCY and uhCG/EGF (Experimental): PTCY for 2 doses on day +3 and +4 after stem cell transplant followed by uhCG/EGF subcutaneously on day +7, +9 and +11 post stem cell transplant
  Interventions: Drug: uhCG/EGF

INTERVENTIONS:
Drug: uhCG/EGF — PTCY for 2 doses on day +3 and +4 after stem cell transplant followed by uhCG/EGF subcutaneously on day +7, +9 and +11 post stem cell transplant

SUMMARY:
So this a Phase I study with primary objective to determine the feasibility and safety of combining post-transplant cyclophosphamide and urinary-derived human chorionic gonadotropin and epidermal growth factor (uhCG/EGF) as graft versus host disease prophylaxis in stem cell transplant with MMUDs Secondary objectives are to determine the incidence acute and chronic GVHD, progression-free survival , and overall survival

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hematologic malignancy who have the indication for Allogeneic SCT and have no MRD or MUD.
2. Age 18-70 years old
3. Performance score of at least 80% by Karnofsky
4. Adequate kidney and liver function as demonstrated by:

   1. Creatinine clearance should be >60 ml/min
   2. Total Bilirubin <1.5, ALT/AST/Alk Phos < 2.5 x normal. No evidence of chronic active hepatitis or cirrhosis.
5. Negative Beta HCG test in a woman with childbearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization. Women of childbearing potential must be willing to use an effective contraceptive measure while on study.
6. Patient or patient's legal representative, parent(s) or guardian able to sign informed consent.

Exclusion Criteria:

1. Positive for HIV, HBsAg, HCV or other viral hepatitis or cirrhosis from any cause
2. Active or prior CNS leukemia, unless in complete remission for at least 2 months.
3. History of serious chronic mental disorder or drug-abuse accompanied by documented problems of compliance with therapeutic programs.
4. Uncontrolled infection
5. Donor specific antibodies
6. Ejection fraction <40% or history of heart failure or cardiovascular disease
7. history thrombosis or current thrombosis, family history of thrombosis, severe obesity, or thrombophilia.
8. Previous history hormone responsive cancer
9. history of seizure
10. history of migraine or severe headache
11. history of asthma
12. history of uterine fibroid

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
MTD | day+30 post SCT
  The maximum tolerated dose
Incidence and severity of dose limiting toxicity (DLTs) | day+30 post SCT
  The overall incidence and severity of DLTs for uhCG/EGF

SECONDARY OUTCOMES:
acute GVHD | till day +100 post SCT
  Cumulative incidence of acute GVHD
Chronic GVHD | one year post SCT
  Cumulative incidence of chronic GVHD
Overall survival | one year post SCT
  Death from any cause will be considered an event. Surviving patients will be censored at the time of last follow up.
Disease free survival | one year
  Survival following allogeneic SCT without relapse or progression. Relapse or progression of disease, or death are considered events

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States